CLINICAL TRIAL: NCT00590161
Title: Treatment Efficacy of Pentoxifylline in Patients With Nonalcoholic Steatohepatitis: A Double-blind Randomized Placebo Controlled Trial
Brief Title: Pentoxifylline in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Claudia Zein, Assistant Clinical Professor, Lerner College of Medicine of Case Western Reserve University, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-1196 CWRU CRU
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-08

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Fatty Liver; Nonalcoholic fatty liver disease (NALFD); NAFLD; Nonalcoholic steatohepatitis (NASH); NASH; pentoxifylline
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pentoxifylline (PTX) 400 mg by mouth (PO) three times daily (TID)
  Interventions: Drug: pentoxifylline (PTX)
- 2 (Placebo Comparator): Placebo three times daily (TID)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pentoxifylline (PTX) — 400 mg PO tid
  Arms: 1
Drug: placebo — placebo tid
  Arms: 2

SUMMARY:
One third of the population in the United States has nonalcoholic fatty liver disease (NAFLD). Nonalcoholic steatohepatitis (NASH), the progressive form of NAFLD, can lead to cirrhosis.Currently, there is no proven therapy for patients with NASH. The investigators core hypothesis is that therapy of patients with NASH with pentoxifylline (PTX) for one year will result in improvement of biochemical parameters of liver disease and hepatic histology. The focus of this proposal is on the effectiveness of pentoxifylline (PTX) in improving laboratory and tissue parameters of liver disease, parameters of insulin-resistance, and levels of cytokines in patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18 to 70 years.
* Liver biopsy compatible with NASH, including presence of steatosis and necroinflammatory activity on liver biopsy done during the prior 6 months to study enrollment
* Daily alcohol intake of <30 g for males and <15 g for females;
* Appropriate exclusion of other liver diseases.
* Patients with diabetes mellitus type 2 diagnosis as defined by a previous diagnosis of DM and current therapy with antidiabetic agents, or by fulfillment of 1997 American Diabetic Association (ADA) criteria, may be included if they fulfill the following criteria: (i) therapeutic regimen limited to specific oral agents including sulfonylureas (e.g. glipizide and glyburide) and/or biguanides (e.g. metformin); (ii) stable therapeutic regimen as defined by no changes in oral agents for at least 3 months; (iii) Hemoglobin A1C (HgbA1C) < 8.5 %.

Exclusion Criteria:

* History of past excessive alcohol drinking (as defined above) for a period longer than 2 years at any time in the past 10 years.
* Current consumption of alcohol >30 g daily for males and >15 g daily for females.
* Positive testing for hepatitis B surface antigen, hepatitis C virus antibody, or ribonucleic acid (RNA) of hepatitis C virus of deoxyribonucleic acid (DNA) of hepatitis B virus.
* Patients taking medications known to cause steatosis.
* Other causes of liver disease suspected by history, family interview, or laboratory testing.
* Patients with cirrhosis defined by stage 4 fibrosis on liver biopsy, or if the patient shows unequivocal clinical evidence of portal hypertension, such as thrombocytopenia, splenomegaly, or esophageal varices.
* Patients taking medications of possible benefit in NASH within 3 months prior to the liver biopsy. These medications include Vitamin E, Betaine, S-adenosylmethionine (SAM-e), thiazolidinediones, and acarbose.
* Patients with diabetes mellitus who are on Insulin therapy.
* Patients with diabetes mellitus on therapy with thiazolidinediones or alpha-glucosidase inhibitors such as acarbose
* Hypersensitivity to pentoxifylline or the methylxanthines (caffeine, theophylline, theobromine).
* History of cerebral or retinal hemorrhage.
* Other medical comorbidities (such as cardiac, central nervous system, renal, cancer) that would interfere with completion of the study.
* Patients taking Theophylline or Coumadin because of potential drug-drug interactions with Pentoxifylline.
* Pregnant or nursing women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia O Zein, MD, MSc, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - Louis Stokes VA Medical Center, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Zein CO, Yerian LM, Gogate P, Lopez R, Kirwan JP, Feldstein AE, McCullough AJ. Pentoxifylline improves nonalcoholic steatohepatitis: a randomized placebo-controlled trial. Hepatology. 2011 Nov;54(5):1610-9. doi: 10.1002/hep.24544. Epub 2011 Aug 24. PMID 21748765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between December 2006 and February 2009 at the Liver Clinics of both participating institutions.
Pre-assignment Details: Patients were randomized in a double-blind fashion. Double blinding was maintained until study completion by all subjects.
Groups:
- Pentoxifylline (PTX) 400 mg PO Three Times Daily (TID): 26 subjects received PTX at dose above for one year
- Placebo TID: 29 subjects received placebo as above for one year
Period: Overall Study
Arm/Group | Pentoxifylline (PTX) 400 mg PO Three Times Daily (TID) | Placebo TID
Started | 26 | 29
Completed | 23 | 26
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pentoxifylline (PTX) 400 mg PO (by Mouth) TID: 26 subjects received PTX at dose above for one year
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline (PTX) 400 mg PO (by Mouth) TID | Placebo TID | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 27 | 50
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 50.5 (12.7) | 49.6 (9.6) | 50 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Histological Improvement of at Least 2 Points in NAFLD Activity Score (NAS) on Liver Biopsy After One Year.
Description: The NAFLD Activity Score (NAS) grades NAFLD on liver biopsy based on the individual scoring of steatosis, inflammation and balloning. The NAS is assessed on a scale of 0 to 8 with higher scores indicating more severe disease and lower scores indicating less severe disease. NAS is obtained by adding steatosis(assessed on a scale of 0 to 3), inflammation (assessed on a scale of 0 to 3) and ballooning (assessed on a scale of 0 to 2).
Time Frame: 1 year (Baseline liver biopsy done at study entry, and subsequent liver biopsy done after one year of therapy with pentoxifylline or placebo)
Population: Intention to treat analysis included all participants and for this analysis patients without available end of study liver biopsy were imputed as treatment failures. Results showed here are continuous variable analysis of NAS score change in patients with available end of study liver biopsy (per protocol analysis)
Measure: Mean (Standard Deviation); unit: NAS score units
Groups:
- Pentoxifylline 400 mg PO Tid: 26 subjects received PTX at dose above for one year
Arm/Group | Pentoxifylline 400 mg PO Tid | Placebo Tid
Number analyzed (Participants) | 20 | 26
NAS score units | -1.6 (1.1) | -0.1 (1.4)

ADVERSE EVENTS:
Arm/Group | Pentoxifylline 400 mg PO Tid | Placebo Tid
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 11/26 | 14/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline 400 mg PO Tid (N=26) | Placebo Tid (N=29)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Bloating (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (General disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lightheadedness (General disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No